CLINICAL TRIAL: NCT02241226
Title: Self-Directed Biological Transformation Initiative
Acronym: SBTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Harvard University (Other); Scripps Translational Science Institute (Other); Duke University (Other); Chopra Center for Wellbeing (Unknown); Mount Sinai Hospital, New York (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Paul J. Mills, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBTI
Record Dates: First submitted 2014-09-09; First posted 2014-09-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Healthy
Keywords: wellbeing; meditation; Ayurveda; yoga; herbs; health; longevity; individuals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perfect health course (Experimental): Perfect health course at the Chopra Center for Wellbeing
  Interventions: Behavioral: Perfect Health Course
- Resort group (No Intervention): Resort group at the La Costa resort

INTERVENTIONS:
Behavioral: Perfect Health Course — The Perfect Health course as taught at the Chopra Center for Wellbeing
  Arms: Perfect health course

SUMMARY:
It is becoming increasingly recognized in the literature that ancient practices for wellbeing, including meditation, yoga, and specific herbs, can improve health and promote longevity. While studies have documented such effects for a variety of individual practices for wellbeing, few studies have taken a more whole systems approach that is simultaneously inclusive of numerous practices. This intervention study, the "Self-Directed Biological Transformation Initiative", will examine the effects of a comprehensive whole systems approach to wellbeing on key biochemical, physiological, and psychosocial endpoints. Participants randomized to the Perfect Health program at the Chopra Center for Wellbeing will be compared to individuals not taking the program.

DETAILED DESCRIPTION:
SPECIFIC AIMS

1. To examine the effects of the Self-Directed Biological Transformation Initiative (SBTI) course participants compared to control group participants on key biochemical and physiological markers.
2. To examine the effects of the SBTI course participants compared to control group participants on short- and long-term changes in heart rate variability, level of activity, and sleep quality.
3. To examine the effects of the SBTI course participants as compared to control group participants on mood and wellbeing.

BACKGROUND AND SIGNIFICANCE It has long been thought that ancient practices can promote longevity and wellbeing but there is little empirical evidence and it is difficult to test this under controlled or experimental conditions. Recently, however, there have been several cellular-based markers that may index rate of biological aging. The rate of telomere shortening, as indexed by change in telomere length and telomerase activity, predicts both cellular and human longevity (Lin et al, 2012). It is related to malleable factors, lifestyle and psychological state (Puterman & Epel, 2012). A secondary measure that shows promise of understanding rate of cellular aging is examination of gene expression, particularly genes related to aging. Preliminary evidence suggests that mind-body practices may slow the rate of cellular aging by improving the telomere/telomerase maintenance system. This has been examined in four small studies so far.

In the first study of its kind, a four month intensive lifestyle modification program, including yoga and group support was associated with an increase in telomerase in 39 men with prostate cancer (in preparation). There was no control group in this study. However, those with the greatest decreases in distressing thoughts about having cancer showed the biggest increases in telomerase activity (Ornish et al, 2008). In a second study, healthy men and women were randomized to a 3-month intensive in-residence meditation group or wait list control group. The researchers examined telomerase only post intervention and found that the meditation group had 30% higher telomerase, and further increases in wellbeing were associated with increases in telomerase (Jacobs et al, 2011). In another study with an active control group, examined 39 elderly high stress dementia caregivers. They randomized half the group to Yoga Nidra, listening to a 15 minute tape each day of Yoga Nidra, which includes instruction on breathing and hand movements and half to a control group which listened to a relaxation tape for 15 minutes each day. Eight weeks later, they found greater telomerase increases in the Yoga Nidra group, and across the sample, decreases in depressive symptoms were associated with increases in telomerase activity (Lavretsky et al, 2013).

Similar studies have reported positive effects of such practices on inflammatory profiles and gene expression (Tang, Ma et al. 2009, Bhasin, Dusek et al. 2013, Saatcioglu 2013). Another well studied parameter for practices such as meditation and yoga is heart rate variability (HRV) as it provides a broad measure of autonomic nervous system activity. Observational studies report HRV to be associated with stress in the workplace,(Jarczok, Jarczok et al. 2013) depressive and anxiety disorders (Gorman and Sloan 2000), and in individuals with chronic somatic complaints (Tak, Riese et al. 2009). Meditation and yoga interventions to improve HRV can lead to improved physiologic and clinical outcomes (Wheat and Larkin 2010, Papp, Lindfors et al. 2013). Other parameters can also be of potential benefit in evaluating an individual's overall wellbeing. For example, sleep duration and quality, as well as general activity levels can both contribute to and reflect overall wellbeing. To date, however, lack of compelling data around objective measures of wellbeing is in large part due to challenges associated with long term monitoring of monitoring of appropriate patient populations. However, recent advances in biosensor technologies have overcome this limitation and now allow for the non-obtrusive and passive monitoring of individuals for long periods of time. These new data streams of real-time physiologic data, couple with sophisticated and individualized data analytics can potentially identify novel measures of individual wellness, which will allow for the development of personalized therapeutic interventions to improve wellbeing.

Overall, while the results of many of the studies of traditional practices are compelling, in reality, and according the more whole system approaches such as Ayurveda and Chines Medicine, traditional practices are rarely practiced singularly, i.e, typically yoga asanas are practiced with meditation as well as a form of pranayama (breathing). With this consideration, few scientific studies have taken a more comprehensive "whole systems" approach that is simultaneously inclusive of numerous practices. Regarding outcomes, this study will take a systems biology approach to examining the biochemical, physiological, and psychosocial effects of the intervention. It is anticipated that the findings will demonstrate the value of taking a more inclusive and comprehensive whole systems approach to improving wellbeing and improved health.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 40-80 years

   Exclusion Criteria:
2. Self-reported diagnosis of a major medical condition, such as cancer (including those who have received past radiation or chemotherapy treatment), heart disease, autoimmune disease, or diabetes, as these can affect the cell aging system and possibly the ability for telomerase to change in short periods
3. Individuals taking antidepressant medication will be excluded since such medication appears to increase telomerase (Wolkowitz et al, 2010)
4. Individuals with diagnosed PTSD will be excluded; there is evidence that those with PTSD may have lower telomere length as compared to those without PTSD (O'Donovan et al, 2011). It is currently unknown how PTSD may impact telomerase levels
5. Estrogen use is excluded as it increases telomerase (Lin et al, 2011)
6. Smokers will be excluded since smoking decreases telomerase. We will base smoking status on self report. If participants have not smoked regularly for the past 6 months, they will be considered a 'non-smoker
7. Pregnant women are excluded since the cell aging system changes during pregnancy in ways that have not been studied
8. Participants with a Body Mass Index (BMI) of 35 or greater will be excluded due to differences in telomerase activity in obese women
9. Potential eligible participants who are unable to secure the week off from work or other responsibilities will not be enrolled
10. Known atrial fibrillation or other chronic dysrhythmia

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in RNA expression | Assessed pre and post 7 day intervention
  Blood samples will be collected for RNA expression and assayed using standardized methodologies
Change in cytokine levels | Assessed pre and post 7 day intervention
  Blood samples will be collected for inflammatory cytokine levels and determined via standardized ELISA methods
Change in telomerase activity | Assessed pre and post 7 day intervention
  Blood samples will be collected for PBMC telomerase activity and assayed using standardized methodologies
Change in neurohormome levels | Assessed pre and post 7 day intervention
  Blood and saliva samples will be collected for neurohormone levels and be determined via standardized ELISA methods

SECONDARY OUTCOMES:
Change in heart rate variability | Assessed pre and post 7 day intervention and one month follow-up
  ECG activity will be obtained via continuous wearable wireless sensor

OTHER OUTCOMES:
Change in quality of life | Assessed pre and post 7 day intervention and one month follow-up
  A set of standardized and validated questionnaires will be administered
Change in gut microbiome populations | Assessed pre and post 7 day intervention and one month follow-up
  Stool samples will be collected to determine gut microbiome using standardized methodologies
Change in mood | Assessed pre and post 7 day intervention and one month follow-up
  A set of standardized and validated questionnaires will be administered
Change in spiritual wellbeing | Assessed pre and post 7 day intervention and one month followup
  A set of standardized and validated questionnaires will be administered

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Mills, PHD, Study Director — University of California, San Diego; Rudolph E Tanzi, PhD, Study Chair — Harvard University; Deepak Chopra, MD, Study Chair — Chopra Center for Wellbeing & University of California, San Diego; Elizabeth Blackburn, PhD, Principal Investigator — University of California, San Francisco; Elissa Epel, PhD, Principal Investigator — University of California, San Francisco; Sheila Patel, MD, Principal Investigator — Chopra Center for Wellbeing & University of California, San Diego; Valencia Porter, MD, Principal Investigator — Chopra Center for Wellbeing & University of California, San Diego; Eric Schadt, PhD, Principal Investigator — MOUNT SINAI HOSPITAL; Steven Steinhubl, MD, Principal Investigator — Scripps Translational Science Institute, Scripps Research Institute; Eric Topel, MD, Principal Investigator — Scripps Translational Science Institute, Scripps Research Institute; Murali Doraiswamy, MD, Principal Investigator — Duke University
Locations (1):
- Chopra Center for Wellbeing, Carlsbad, California, United States